CLINICAL TRIAL: NCT04854798
Title: Ultrasound Neural and Immunomodulation Treatment Evaluation Study (UMN-SW) for COVID-19 With Wearable Ultrasound Device
Brief Title: UNITE Study (UMN-SW) for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: SecondWave Systems Inc. (Industry); DARPA (United States Department of Defense) (Unknown); MCDC (United States Department of Defense) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00050829
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Covid19; Cytokine Storm; Inflammation
Keywords: Covid19; Cytokine Storm; Inflammation
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Inflammation

STUDY DESIGN:
Intervention Model Description: The participants will be randomized to two groups: ultrasound group and control group. All participants will still receive standard clinical care. The ultrasound group will receive daily ultrasound application to the spleen for up to 7 days, in addition to the standard clinical care. The control group will receive standard clinical care without ultrasound stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Group (Experimental): Daily ultrasound application to the spleen of approximately 18 minutes for up to 7 days, in addition to standard clinical care.
  Interventions: Device: Splenic Ultrasound
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Device: Splenic Ultrasound — Daily ultrasound application to the spleen of approximately 18 minutes for up to 7 days, in addition to standard clinical care
  Other Names: SecondWave Systems investigational MINI device
  Arms: Ultrasound Group

SUMMARY:
The research objective of the UNITE Study is to assess device feasibility of ultrasound application to the spleen using a small wearable ultrasound system to assess its effect on coronavirus disease 2019 (COVID-19) in a pilot study using an early stage prototype device.

Specific Aims:

1. Determine the feasibility of splenic ultrasound with a prototype wearable device in affecting physiological markers in COVID-19 infected patients between an ultrasound group versus a control group for the primary analyses; and
2. Evaluate the potential capabilities of splenic ultrasound with this prototype wearable device in affecting additional outcomes in COVID-19 infected patients in the ultrasound group compared to a control group.

DETAILED DESCRIPTION:
Ultrasound is widely used in human medicine because it is safe, non-invasive, and painless. The same kind of ultrasound that is used for imaging (for example, to visualize babies in utero) may be able to treat inflammatory diseases including COVID-19. COVID-19 is a disease caused by infection with the SARS-CoV-2 virus. Some COVID-19 patients develop a severe respiratory disease called acute respiratory distress syndrome and this disease is caused, in part, by a significant increase in inflammatory factors. Clinical therapies that reduce this elevated inflammation in the body (e.g., inflammation molecules in your body called cytokines) may be capable of diminishing symptoms in severe cases of COVID-19.

Multiple studies in animals with hyper-inflammation conditions (e.g., inflammatory arthritis and sepsis/LPS injections) and recent human studies (e.g., for the treatment of joint inflammation in Rheumatoid Arthritis) have shown that ultrasound applied to the spleen can suppress blood/genetic markers of inflammation. Similar inflammatory markers, or cytokines, are elevated in the lungs of COVID-19 patients and believed to cause severe symptoms. Splenic ultrasound can potentially lower these inflammatory cytokines without hindering antibody production, leading to clinical improvements in COVID-19 patients.

This study will employ investigational ultrasound devices produced by SecondWave Systems called the MINI (Miniature Immunotherapy and Neuromodulation Instrument).

There will be two groups in this study with 29 participants in each group. One group will receive ultrasound application to the spleen, in addition to the standard clinical care. A control group will receive standard clinical care without splenic ultrasound. Each ultrasound application session will last about 30 minutes per day for 7 days, unless the participant is discharged sooner. For ultrasound stimulation, a small wearable ultrasound device is positioned on the upper left abdomen area over the ribs. The ultrasound session on the first study day includes a period of 5-10 minutes when study personnel use an ultrasound imaging device to locate the spleen and to position the wearable MINI device in a proper location around the ribs area. Daily stimulation consists of an approximately 18-minute period for application of ultrasound to the spleen. Collection of clinical outcome data and daily blood draws will be performed in each participant throughout the study through Day 8. Additional data collected from each participant during their routine clinical care beyond their study involvement will also be analyzed together with the study data to evaluate the specific aims of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Positive for SARS-CoV-2 (via PCR)
* Decreased blood oxygen saturation: Room air SaO2 < 94% and/or requiring supplemental oxygen at a flow rate of 2 L/min or greater
* Admission to the hospital

Exclusion Criteria:

* Pregnant women
* Asplenia
* Ascites
* Open wound/sores near the stimulation site
* Recent abdominal surgery
* Splenomegaly
* Mechanically ventilated (if patient goes onto mechanical ventilation while participating in the study, they can continue ultrasound treatment if recommended by SOC clinician and investigators of this study)
* Comfort care status
* Any other clinical reasons deemed by the investigators of the study in which the patient would not be an appropriate candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
IL-6 levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Percentage of participants with observed change in IL-6 levels
IL-1β levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Percentage of participants with observed change in IL-1β levels

SECONDARY OUTCOMES:
Hospitalized days based on the ordinal scale | Baseline to date of recovery, assessed up to 14 days
  Mean change in the number of days of hospitalized state of patients (based on the ordinal scale) in the ultrasound group versus the control group

OTHER OUTCOMES:
Ordinal scale values over time | Baseline to Day 8 (end of stimulation; last observation carried forward if date of discharge or death is earlier)
  Between-arm comparison of area under the curve of ordinal scale values (absolute and normalized) from baseline to end of treatment between groups.
CRP levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Change in CRP levels
Hypoxemia duration | Baseline to date of discharge or date of death, whichever came first, assessed up to 6 months
  Change in duration of hypoxemia
D-dimer levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Change in D-dimer levels
Mechanical ventilation | Baseline to date of discharge or date of death, whichever came first, assessed up to 6 months
  Change in rate of requiring mechanical ventilation
Mortality rate | Baseline to date of discharge or date of death, whichever came first, assessed up to 6 months
  Change in mortality rate
TNF levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Change in serum cytokine concentration of TNF
IL-10 levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Change in serum cytokine concentration of IL-10
IFN-gamma levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Change in serum cytokine concentration of IFN-gamma
IL-18 levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Change in serum cytokine concentration of IL-18
IL2R-alpha levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Change in serum cytokine concentration of IL2R-alpha
IL-4 levels | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Change in serum cytokine concentration of IL-4
RNAseq pathways | Baseline to Day 8 (end of stimulation; or date of discharge or death if earlier)
  Change in RNAseq identified pro-inflammatory pathways

CONTACTS AND LOCATIONS:
Overall Officials: Erik Peterson, M.D., Principal Investigator — University of Minnesota; Andrew Olson, M.D., Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - M Health Fairview Ridges Hospital, Burnsville, Minnesota
  - M Health Fairview St. Joseph's Hospital, Saint Paul, Minnesota

REFERENCES:
- See also: First-in-human demonstration of splenic ultrasound stimulation for non-invasively controlling inflammation — https://www.medrxiv.org/content/10.1101/2020.07.14.20153528v2